CLINICAL TRIAL: NCT02612363
Title: The Effect of Early Goal Directed Sedation on Microcirculation in Septic Shock Patients With Mechanical Ventilation
Brief Title: Early Goal Directed Sedation on Microcirculation in Septic Shock
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015ZDSYLL016.0
Record Dates: First submitted 2014-10-28; First posted 2015-11-23 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Septic Shock
Keywords: septic shock; sedation; microcirculation
MeSH Terms: conditions — Shock, Septic | interventions — Dexmedetomidine; Drug and Narcotic Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early goal directed sedation group (Experimental): Dexmedetomidine for sedation in early goal directed sedation group
  * Analgesia
  * Dexmedetomidine start at 0.7ug/kg/hour
  * Dose range: 0.2- 0.7 u/kg/hour
  * Supplemental other sedatives at lowest effective dose Target Richmond Agitation-Sedation Scale score of -2 to +1 to achieve sedation goal in EGDS group
  Interventions: Drug: Dexmedetomidine for sedation
- Standard sedation (Placebo Comparator): Control drug for sedation in early goal directed sedation group
  * Analgesia
  * Control drug
  * Supplemental other sedatives at lowest effective dose for standard sedation Target Richmond Agitation-Sedation Scale score of -2 to +1 to achieve sedation goal
  Interventions: Drug: Dexmedetomidine for sedation

INTERVENTIONS:
Drug: Dexmedetomidine for sedation — Dexmedetomidine or control drug for sedation
  * Analgesia
  * Propofol at lowest dosage.
  * Dose range: 0.1- 0.7 u/kg/hour
  * Target RASS score of -2 to +1
  * Supplemental other sedatives at lowest effective dose
  Other Names: Control drug for sedation

SUMMARY:
The investigators will conduct a prospective, single-center, randomized, double-blinded, controlled study to investigate the effect of early goal directed sedation on microcirculation in early septic shock patients.

DETAILED DESCRIPTION:
Recent studies suggest that early goal directed sedation might improve the outcome of critically ill patients. The investigators will conduct a prospective, single-center, randomized, double-blinded, controlled study to investigate the effect of early goal directed sedation on microcirculation in early septic shock patients with relative stable hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock patients despite early goal directed therapy
* Required sedation

Exclusion Criteria:

* Age< 18
* Pregnancy
* Bradycardia (HR<55bpm)
* Systolic blood pressure < 80 mmHg / mean arterial pressure < 50 mmHg on maximal support
* Death imminent
* Unlikely to survive 90 days
* Acute liver failure
* Dementia
* High-grade block in the absence of a functioning pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Microcirculatory function as assessed by perfused vessel density | one hour
  Microcirculatory parameter

SECONDARY OUTCOMES:
Dose of sedatives and analgesic agents | 14 days
Oxygen metabolic: lactate clearance time | six hours

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, Ph.D., Principal Investigator — Southeast University
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided